CLINICAL TRIAL: NCT01011153
Title: Comparison of Diagnostic and Biopsy/Referral Sensitivity to Melanoma Between Three Groups of Physicians and MelaFind
Brief Title: Survey Study - Sensitivity Comparison Between MelaFind and Physician Group
Status: Completed | Type: Observational
Sponsor: MELA Sciences, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20063
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Results first posted 2011-01-24 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Dermatologists

SUMMARY:
This survey study purposes to determine and compare the biopsy/referral sensitivity and specificity of MelaFind to the average biopsy/referral sensitivity and specificity of dermatologists. 241 subjects logged into system but only 183 signed consents and completed the intake survey. Out of these 183, 155 were accounted for in the data analysis after exclusions were removed from the pool of subjects.

DETAILED DESCRIPTION:
Early detection of melanoma is critical for favorable prognosis, since patients with earlier stage melanomas have a much higher probability of survival than with later stages. The traditional method of early detection has been with serial total body skin exams where the health care provider examines all skin surfaces, including mucosa, for suspicious pigmented lesions. Studies have demonstrated that the diagnostic accuracy of physicians for melanoma depends on the level of dermatological training. More important than being able to make a diagnosis of melanoma on clinical impression is the ability to make an appropriate decision to biopsy the lesion. Primary care physicians (PCPs) are often expected to screen for melanoma and only refer to dermatologists when there is a high clinical suspicion of melanoma. However, if PCPs are not adept at diagnosing melanoma, then opportunities for early diagnosis and treatment could be missed. Conversely, the morphology of benign pigmented lesions can often mimic that of early melanomas, resulting in potentially unnecessary dermatology referrals, biopsies, and patient anxiety. Studies have indicated that there is great variability in the ability of PCPs to make a correct decision to biopsy/refer a pigmented lesion (1.5 times greater than dermatologists) as well as for diagnosing melanoma (over 2.5 times greater than dermatologists). To aid in detection of early melanomas, new technologies are being developed.

One such technology is MelaFind, an investigational device that has been developed to give a recommendation for biopsy (or not) of pigmented skin lesions to rule out melanoma. Our hypothesis is that MelaFind will have equal or better sensitivity than pigmented lesion experts in making an appropriate recommendation for biopsy (i.e., MelaFind will be at least as accurate as dermatologists in recommending biopsy for melanomas).

ELIGIBILITY:
Inclusion Criteria:

* Board Certified physicians or equivalent

Exclusion Criteria:

* Did not participate in EOS Protocols 20061 or 20081

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Three groups of health care providers who commonly encounter the skin will participate in the study. The population will comprise ninety physicians of which thirty are pigmented skin lesions experts, thirty general dermatologists and thirty primary care physicians.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suephy Chen, MD, Principal Investigator — Emory University

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Physicians were selected from the membership list of the AAD and lists provided by SK&A Healthcare Information Solutions. A letter was then sent inviting them to participate. For each who replied positively,an access code was mailed with which to log on to the study. 241 subjects logged into system,183 signed consents & completed the Intake Survey.
Pre-assignment Details: Participants were grouped according to responses to an Intake Survey, completed after Consent and before reading any study cases. A maximum of 130 cases were reviewed,each one consisting of 3 clinical images and a case history. MelaFind results were not provided as part of each case and were only used for sensitivity and specificity calculations.
Groups:
- General Dermatologists: Dermatologists were defined as board-certified dermatologists who did not participate in previous EOS Protocols 20061 and 20081
- Pigmented Skin Lesion Experts: Pigmented Skin Lesion Expert were defined as board-certified dermatologists who spend at least 25% of their practice time evaluating pigmented skin lesions (PSLs)
- Primary Care Physicians: Primary Care Physicians(PCPs) were defined as physicians who deliver primary care service to adult patients (e.g., internists, general practitioners, family practitioners, and geriatricians).
Period: Overall Study
Arm/Group | General Dermatologists | Pigmented Skin Lesion Experts | Primary Care Physicians
Started | 54 | 75 | 54
Completed | 46 | 64 | 45
Not Completed | 8 | 11 | 9
Not completed — Less than 78 cases completed | 8 | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Dermatologists | Pigmented Skin Lesion Experts | Primary Care Physicians | Total
Number analyzed (Participants) | 54 | 75 | 54 | 183
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 54 | 75 | 54 | 183
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Female | 16 | 36 | 23 | 75
  Male | 32 | 35 | 26 | 93
  Unknown | 6 | 4 | 5 | 15
Region of Enrollment [Number; unit: participants]
  United States | 54 | 75 | 54 | 183

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Biopsy/Referral Sensitivity of MelaFind and Dermatologists (Pigmented Skin Lesion Experts and General Dermatologists)
Description: Sensitivity is the proportion of positive cases (i.e., histologically confirmed melanoma) identified as positive. Specificity is the proportion of negative cases (i.e., histologically confirmed non-melanoma) identified as negative. Because the number of cases given to each dermatologist varied, both sensitivity and specificity were computed for each dermatologist. The primary outcome as stated was to compare the sensitivity and specificity of all dermatologists to that of MelaFind. These metrics, for both the dermatologists and MelaFind, were calculated based on the same 130 lesions.
Time Frame: April 2010
Population: Participants were invited to enroll in this study via mail. Minimum number of participants was determined by statistician based on power analyses and number of cases completed. The time frame of the study was about 6 months and the comparison between Dermatologists and MelaFind is presented in the statistical analysis section below.
Measure: Mean (95% Confidence Interval); unit: Proportion of True Cases
Groups:
- Dermatologists: Dermatologists were defined as board-certified dermatologists who were General Dermatologists and Pigmented Skin Lesion Experts, according to the Intake Survey. Dermatologists in this group did not participate in previous EOS Protocols 20061 and 20081. Each dermatologist was given up to 130 cases (each one consisting of 3 clinical images and a case history) consistinf of 65 positive cases (i.e., histologically confirmed melanoma) and 65 negative cases (i.e., histologically confirmed non-melanoma)
- MelaFind: MelaFind imaged 130 cases which consisted of 65 positive cases (i.e., histolgoically confirmed melanoma) and 65 negative cases (i.e., histologically confirmed non-melanoma).
Arm/Group | Dermatologists | MelaFind
Number analyzed (Participants) | 110 | 1
Proportion of True Cases
  Proportion of True Positive Cases (Sensitivity) | 0.72 (8.4) [0.66 to 0.78] | 0.97 (0) [0.9 to 0.99]
  Proportion of True Negative Cases (Specificity) | 0.51 (0) [0.43 to 0.58] | 0.09 (0) [0.04 to 0.19]
Statistical Analysis 1: Comparison: Dermatologists vs MelaFind; Using True Positives/All Positives, sensitivity values were calculated for MelaFind as well as the average of the 110 dermatologists; Test type: Non-Inferiority or Equivalence — Sample sizes computed based on data from smaller studies provided 90% power for the comparison of sensitivity. Under the alternative hypothesis that the biopsy sensitivity of MelaFind would be 0.10 greater than the average biopsy/referral sensitivity of physicians (combined or separate), the probability that a 95% CI lies entirely above zero will be at least 90% when the standard error of the estimated difference is at most 0.0308; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [0.18 to 0.32], Standard Deviation 0.03

2. Secondary Outcome: Comparison of Biopsy/Referral Sensitivity and Specificity of MelaFind to the Average of Biopsy/Referral Sensitivity & Specificity in Each of the Three Groups of Physicians: Pigmented Skin Lesion Experts, General Dermatologists, and Primary Care Physicians
Description: Sensitivity is the proportion of positive cases (i.e., histologically confirmed melanoma) identified as positive. Specificity is the proportion of negative cases (i.e., histologically confirmed non-melanoma) identified as negative. Because the number of cases given to each dermatologist varied, both sensitivity and specificity were computed for each dermatologist. The primary outcome as stated was to compare the sensitivity and specificity of each group of physicians to that of Melafind, which is presented in the statistical analysis.
Time Frame: December 2009
Population: Each category was diminished after excluded subjects were taken into account. These included subjects who did not complete at least 78 cases, subjects who previously participated in other EOS studies, pediatricians, and a board eligible dermatologist.
Measure: Mean (95% Confidence Interval); unit: Proportion of True Cases
Groups:
- General Dermatologists: General Dermatologists were defined as board-certified dermatologists who did not participate in previous EOS Protocols 20061 and 20081. Each dermatologist was given up to 130 cases (each one consisting of 3 clinical images and a case history) consisting of 65 positive cases (i.e., histologically confirmed melanoma) and 65 negative cases (i.e., histologically confirmed non-melanoma)
- Pigmented Skin Lesion Experts: Physicians who spend at least 25% of their practice time examining pigmented skin lesions. Each PSL Expert was given up to 130 cases (each one consisting of 3 clinical images and a case history) consisting of 65 positive cases (i.e., histologically confirmed melanoma) and 65 negative cases (i.e., histologically confirmed non-melanoma).
- Primary Care Physicians: Physicians who are not Board Certified Dermatologists and Pediatricians. Each PCP was given up to 130 cases (each one consisting of 3 clinical images and a case history) consisting of 65 positive cases (i.e., histologically confirmed melanoma) and 65 negative cases (i.e., histologically confirmed non-melanoma).
- MelaFind: MelaFind imaged the 130 cases, the 65 positive cases (i.e., histologically confirmed melanoma) and the 65 negative cases (i.e., histologically confirmed non-melanoma). Sensitivity was calculated based on the correct identification of the 65 positive cases and specificity was calculated based on the correct identification of the 65 negative cases.
Arm/Group | General Dermatologists | Pigmented Skin Lesion Experts | Primary Care Physicians | MelaFind
Number analyzed (Participants) | 46 | 64 | 45 | 1
Proportion of True Cases
  Proportion of True Positive Cases (Sensitivity) | 0.73 (8.7) [0.67 to 0.80] | 0.71 (8.1) [0.65 to 0.77] | 0.71 (10.9) [0.64 to 0.78] | 0.97 (0) [0.90 to 0.99]
  Proportion of True Negative Cases (Specificity) | 0.51 (0) [0.43 to 0.60] | 0.50 (0) [0.42 to 0.58] | 0.45 (0) [0.37 to 0.53] | 0.09 (0) [0.04 to 0.19]
Statistical Analysis 1: Comparison: Primary Care Physicians vs MelaFind; Sensitivity; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [0.19 to 0.34], Standard Deviation 0.04
Statistical Analysis 2: Comparison: General Dermatologists vs MelaFind; Sensitivity; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.24, 95% CI 2-sided [0.16 to 0.31], Standard Deviation 0.04
Statistical Analysis 3: Comparison: Pigmented Skin Lesion Experts vs MelaFind; Sensitivity; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.26, 95% CI 2-sided [0.19 to 0.33], Standard Deviation 0.03
Statistical Analysis 4: Comparison: Primary Care Physicians vs MelaFind; Specificity; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.46 to -0.25], Standard Deviation 0.05
Statistical Analysis 5: Comparison: General Dermatologists vs MelaFind; Specificity; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = -0.42, 95% CI 2-sided [-0.53 to -0.31], Standard Deviation 0.05
Statistical Analysis 6: Comparison: Pigmented Skin Lesion Experts vs MelaFind; Specificity; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.51 to -0.30], Standard Deviation 0.05

3. Secondary Outcome: Determine the Interobserver Variability in Each of the Above Metrics Within Each of the Caregiver Groups.
Description: Each physician was given up to 130 cases and asked whether or not they would biopsy the lesion. Interobserver variability was measured via the kappa statistic indicating how well the physicians' answers to that question agreed within each group. Kappa statistics are reported in the statistical analysis. while numbers rep, they dont reflect the sgreement among the subjects
Time Frame: December 2009
Population: The statistical analysis section contains the Kappa results within Each of the Caregiver Groups
Measure: Number; unit: Number of Cases
Groups:
- Dermatologists: General Dermatologists were defined as board-certified dermatologists who did not participate in previous EOS Protocols 20061 and 20081. Each dermatologist was given up to 130 cases (each one consisting of 3 clinical images and a case history) consisting of 65 positive cases (i.e., histologically confirmed melanoma) and 65 negative cases (i.e., histologically confirmed non-melanoma)
- All Partipants: All Participants are the General Dermatologists, Pigmented Skin Lesion Experts and Primary Care Physicians combined.
Arm/Group | Dermatologists | Pigmented Skin Lesion Experts | Primary Care Physicians | All Partipants
Number analyzed (Participants) | 46 | 64 | 45 | 155
Number of Cases | 5927 | 8263 | 5844 | 20034
Statistical Analysis 1: Comparison: Dermatologists; Test type: Superiority or Other; ANOVA — No comparison is being made; Kappa = 0.313, Standard Error of Mean 0.003 — There is no threshold level-this is a measurement of variability among responses provided by the participants
Statistical Analysis 2: Comparison: Pigmented Skin Lesion Experts; Test type: Superiority or Other; ANOVA — No comparison is being made; Kappa = 0.276, Standard Error of Mean 0.002 — There is no threshold level-this is a measurement of variability among responses provided by the participants
Statistical Analysis 3: Comparison: Primary Care Physicians; Test type: Superiority or Other; ANOVA — No comparison is being made; Kappa = 0.200, Standard Error of Mean 0.003 — There is no threshold level-this is a measurement of variability among responses provided by the participants
Statistical Analysis 4: Comparison: All Partipants; Test type: Superiority or Other; ANOVA — N/A - No comparison is being made; Kappa = 0.256, Standard Error of Mean 0.001 — There is no threshold level-this is a measurement of variability among responses provided by the participants

4. Secondary Outcome: To Compare Biopsy/Referral Performance and Diagnostic Performance Using Areas Under the Corresponding Receiver Operating Characteristic (ROC) Curves That Illustrate the Trade-offs Between Sensitivity and Specificity Between Three Groups of Physicians.
Description: For each case reviewed, physicians were asked if they thought the lesion was a melanoma (diagnostic sensitivity/specificity) and whether or not they would biopsy or refer the lesion (biopsy/referral sensitivity/specificity. These measurements were compared using areas under the corresponding receiver operating characteristic curves. (see statistical analysis for results) ROC curves (reciver operating curves) are plotted on graphs with an x-axis of sensitivity and a y-axis of 1-specificity.
Time Frame: June 2010
Measure: Geometric Mean (Standard Deviation); unit: Area Under Curve for biopsy/referral
Arm/Group | General Dermatologists | Pigmented Skin Lesion Experts | Primary Care Physicians
Number analyzed (Participants) | 46 | 64 | 45
Area Under Curve for biopsy/referral
  Area Under Curve for Biopsy/Referral | 0.65 (0.03) | 0.63 (0.03) | 0.59 (0.02)
  Area Under Curve for Diagnostic | 0.68 (0.03) | 0.66 (0.03) | 0.61 (0.03)

ADVERSE EVENTS:
Description: No safety analyses were planned for this survey study which used cases in which medical management had already been planned and carried out.
Arm/Group | General Dermatologists | Pigmented Skin Lesion Experts | Primary Care Physicians
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The only limitation to having complete data sets was the time a physician was willing to spend on completing the survey.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days